CLINICAL TRIAL: NCT06215300
Title: The Effect of Polymorphism of the GUCY1A3 rs7692387 Gene on Cardiovascular Events After Coronary Artery Bypass Grafting.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Novosibirsk Scientific Research Institute for Circulatory Pathology (Other)
Responsible Party: Sponsor
Other Study IDs: GUCY1A3 rs7692387
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: to Evaluate the Association of GUCY1A3 rs7692387 Gene Polymorphism Carrier on the Development of Cardiovascular Events After Coronary Artery Bypass Grafting
Keywords: cardiovascular system, coronary artery bypass grafting, aspirin resistance, GUCY1A3 gene polymorphism rs7692387, soluble guanylate cyclase (rGC)
MeSH Terms: interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- genotype GG: GG
  Interventions: Genetic: coronary artery bypass grafting
- genotype AG/АА: AG/АА
  Interventions: Genetic: coronary artery bypass grafting

INTERVENTIONS:
Genetic: coronary artery bypass grafting — coronary artery bypass grafting

SUMMARY:
Polymorphism in the GUCY1A3 gene worsens the activity of rCC, causing vasoconstriction and increased platelet aggregation. Studies have shown the association of the GUCY1A3 gene with the risk of coronary heart disease and its complications, with ischemic stroke

DETAILED DESCRIPTION:
Acetylsalicylic acid is indicated for the prevention of cardiovascular complications after CABG. Class I. The level of evidence A. ECS recommendations, Russian recommendations of cardiologists. However, the main problem of CABG remains thrombotic and thromboembolic complications in the immediate and long-term postoperative period, despite taking acetylsalicylic acid. According to various sources, the resistance to ASA among the population ranges from 5 to 45%. Resistance to ASA is primarily associated with genetic factors: the presence of polymorphisms of genes encoding platelet receptor proteins, and the functional activity of soluble guanylate cyclase (rCC), the synthesis of which is controlled by the GUCY1A3 gene. Studies have shown a link between the GUCY1A3 gene and the risk of coronary heart disease and its complications. The presence of polymorphism in the GUCY1A3 gene significantly worsens the activity of rCC, causing vasoconstriction and increased platelet aggregation. At the same time, acetylsalicylic acid cannot provide effective prevention of thrombotic and thromboembolic complications.

ELIGIBILITY:
Inclusion Criteria:

* Stable ischemic disease 2- 4
* CABG

Exclusion Criteria:

* the need to take any anticoagulants
* thrombocytopenia
* allergy to aspirin.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with IHD
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
myocardial infarction, acute cerebrovascular accident, death from cardiovascular causes. | 12 months
  myocardial infarction, acute cerebrovascular accident, death from cardiovascular causes.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Novosibirsk research institute of circulation pathology, Novosibirsk, Novosibirsk Oblast
  - Aleksey, Novosibirsk